CLINICAL TRIAL: NCT02921776
Title: Improving Outcomes for Mechanically Ventilated Patients With the Digital EZ Board
Brief Title: Vidatalk Communication Application: Usability, Acceptability and Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Vidatak, LLC (Industry)
Responsible Party: Principal Investigator, Mary Beth Happ, Associate Dean for Research and Innovation, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016H0006
Record Dates: First submitted 2016-09-07; First posted 2016-10-03 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Nonverbal Communication; Critical Illness
Keywords: Vidatalk; App; Augmentative and Alternative Communication; iPad; Android; Mechanical ventilation; Patient Communication; Critical Illness
MeSH Terms: conditions — Nonverbal Communication; Critical Illness; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Aim 1- VidaTalk post-extubation (Experimental): Aim 1 is a two group iterative design preliminary to clinical trial. Group 1 and Group 2 will each consist of five previously mechanically ventilated patients who will be recruited from the ICUs at the OSUWMC (Ohio State University Wexner Medical Center), including discharged patients.
  Group 1 will use an initial android prototype of VidaTalk tablet application to be assessed for functionality (ergonomics, ease of use, ease of learning, simplicity, effectiveness and user interface) and usability on customizable communication, picture symbols, and integration with mobile communication devices.
  Group 2 will use an improved alpha prototype of VidaTalk tablet application version engineered from observations made during Group 1 sessions.
  Interventions: Other: Aim 1 - VidaTalk - post-extubation
- Aim 2 - VidaTalk intubated (Experimental): Usability testing preliminary to Clinical Trial (Aim 3). Mechanically Ventilated patients will provide feedback on acceptability, will perform test messages with minimal errors, and will rate VidaTalk an overall average score of 4.5 or higher (Likert-type scale; 1 to 7) on usability questions. Prior to implementing these procedures, the company will perform further iterative design assessments and engineer a Vidatalk tablet application prototype. This prototype will be used with a final group of ten (10) intubated patients receiving mechanical ventilation support to field-test the prototype for functionality (human-device interaction factors, feasibility, and usability) and acceptability.
  Intervention is usability tasks with the VidaTalk app
  Interventions: Other: Aim 2 - VidaTalk - intubated
- Aim 3 - VidaTalk tablet app (Experimental): Test the clinical efficacy of VidaTalk with MV patients by examining qualitative and quantitative endpoints in a clinical setting. 35 intubated patients (oral endotracheal tube or tracheostomy) will be randomized to the intervention arm and will receive a protocolized instruction in the use of the VidaTalk application including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 minutes) each day to check user needs and concerns and will review or retrain on message options if needed.
  Intervention will be receipt of VidaTalk tablet application.
  Interventions: Device: Aim 3 - VidaTalk tablet app
- Aim 3 - attention-control (Other): 35 intubated patients (oral endotracheal tube or tracheostomy) will receive the standard of care, which may include primarily writing tools (paper and pen) and, occasionally, picture or alphabet communication charts.
  Patients randomized to the control group will receive a protocolized introduction to the bedside Android device without the VidaTalk application, focusing instead on a common tablet application. Daily visits will be conducted with control group patients to query on use of the attention-control tablet.
  Interventions will be Aim 3 - attention-control with non-VidaTalk tablet.
  Interventions: Other: Aim 3 - attention-control with non-VidaTalk tablet
- Aim 5-VidaTalk Efficacy in Family caregivers (No Intervention): Aim 5 will test the preliminary efficacy of VidaTalk compared to attention control (AC) on anxiety and depression symptoms in family caregivers during the ICU stay and post-discharge (1-mos; 3-mos; 6-mos) and PTSD-related symptoms post-discharge both qualitatively and quantitatively.
  Aim 5.a.) Psychological outcomes (anxiety, depression, and PTSD-related symptoms) between the two groups will be compared at each time point and across time. Aim 5.b.) Family caregivers' perceived communication difficulty will be measured .Aim 5.c.) Family caregivers' experience of communication while they were visiting the patient who received the VidaTalk app in the ICU and their emotional reactions to communication with a patient will be measured.

INTERVENTIONS:
Other: Aim 1 - VidaTalk - post-extubation — Observation of task completion will be made while patients complete a series of messages using the VidaTalk app:
  * Tell me you are tired
  * Tell me you are having pain
  * Rate this pain
  * Tell me there is pain in your back
  * Tell me your pain is sharp
  * Ask to see the doctor
  * Write your favorite color by drawing with your finger
  * Type "How are you?" Patients will also complete a 1-item difficulty rating and a 3-item After-Scenario Questionnaire (ASQ) after each task.
  Patients will also be asked to (a) comment on the customization of the app and make suggestions; (b) rate the extent to which they would use the device if they were an ICU patient and unable to speak.
  Group 1 only:
  Patients will be asked about their preferences for customizing the VidaTalk app.
  Arms: Aim 1- VidaTalk post-extubation
Other: Aim 2 - VidaTalk - intubated — Usability testing prior to clinical trial. The company will have performed further iterative design assessments and engineered a Vidatalk tablet application prototype for a field-test for functionality (human-device interaction factors, feasibility, and usability) and acceptability. Data will be collected by a trained data collector as in Aim 1 with the addition of Ease of Communication and Frustration ratings before and after the testing sequence. To reduce burden, patients in this group will complete the 3-item ASQ one time after all tasks are completed. They will also complete a 13-item System Usability Scale (SUS).
  Arms: Aim 2 - VidaTalk intubated
Device: Aim 3 - VidaTalk tablet app — Patients in the intervention group will receive a protocolized instruction in the use of the VidaTalk application and mounting of the device including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 minutes) each day to check user needs and concerns and will review or retrain on message options if needed.
  Arms: Aim 3 - VidaTalk tablet app
Other: Aim 3 - attention-control with non-VidaTalk tablet — Patents randomized to the control group will receive a protocolized introduction to the bedside Android device without the VidaTalk app, focusing instead on a common tablet application. Daily visits will be conducted with control group patients to query on use of the attention-control tablet.
  Arms: Aim 3 - attention-control

SUMMARY:
This Phase II Small Business Technology Transfer Research (STTR) will deliver a comprehensive patient communication solution for communication-impaired patients in the intensive care unit that may help decrease days in delirium, decrease anxiety levels, and reduce sedation exposure which are proximal outcomes known to be associated with decreased mechanical ventilation days, shorter lengths of ICU and hospital stay, and lower healthcare cost. The primary goal of this Phase II STTR proposal is to further define user requirements and product specifications and develop a prototype of VidaTalk, a patient-centric, touch pad communication software, to provide mechanically ventilated (MV) patients an evidence-based solution for effectively communicating their needs to care providers and family. A secondary goal is to test the impact of the VidaTalk on clinical outcomes. This study will use mixed methods including observations and interaction with hospitalized patients as they use the VidaTalk tool, surveys and medical record data extraction, product evaluation and brief interview, satisfaction surveys with family members of ICU patients, and focus groups with Registered Nurses.

Specific Aim 1. Develop a commercial prototype of VidaTalk that will include multilingual and customizable messages, compatibility with tablet devices, picture symbols, and integration with mobile communication devices.

Specific Aim 2. Demonstrate usability with iterative user assessment testing in a clinical setting.

Specific Aim 3. Test the clinical efficacy of VidaTalk via android application with MV patients by examining qualitative and quantitative endpoints in a clinical setting. Aim 3 hypothesis: MV patients using VidaTalk will demonstrate significant reductions in patient-reported communication difficulty and frustration, anxiety, sedation exposure, delirium/coma-free days, and improved patient and family satisfaction with ICU care compared to MV patients receiving attention-control (i.e., tablets with health education application).

Specific Aim 4. Validation of electronic visual analogue scale, versus current standard paper scale.

Specific Aim 5 a, b and c. Test the effect of the communication tablet (VidaTalk) on psychological symptoms in family caregivers.

DETAILED DESCRIPTION:
Treatment-induced communication impairment is one of the most common and distressful symptoms to mechanically ventilated intensive care unit (ICU) patients and is associated with anxiety, panic, anger, frustration, sleeplessness, and distress.This Phase II Small Business Technology Transfer Research (STTR) will deliver a comprehensive solution that may help decrease days in delirium, decrease anxiety levels, and reduce sedation exposure which are proximal outcomes known to be associated with decreased mechanical ventilation days, shorter lengths of ICU and hospital stay, and lower healthcare cost. The primary goal of this Phase II STTR proposal is to further define user requirements and product specifications and develop a prototype of VidaTalk (previously TouchTalk), a patient-centric, touch pad communication software, to provide mechanically ventilated (MV) patients an evidence-based solution for effectively communicating their needs to care providers and family. A secondary goal is to test the impact of the VidaTalk on clinical outcomes (e.g., patient-reported communication difficulty and frustration, anxiety, sedation exposure, delirium/coma-free days, and improved patient and family satisfaction with ICU care). This study will use mixed methods including observations and interaction with hospitalized patients as they use the VidaTalk communication tool, surveys and medical record data extraction, product evaluation and brief interview, satisfaction survey with family members of ICU patients and focus groups with Registered Nurses. Our Phase I STTR successfully delivered a beta prototype that met technical feasibility criteria; however, additional requirements emerged as a common theme from user testing and market analysis. The current study will meet the identified needs for VidaTalk to operate on android devices, be customizable to patients' unique message needs, use pictures symbols for communication, and be able to route patient requests to providers who are not present at the bedside.

Specific Aim 1 (Preliminary to Clinical Trial). Develop a commercial prototype of VidaTalk that will include multilingual and customizable messages, compatibility with tablet devices, picture symbols, and integration with mobile communication devices.

Specific Aim 2 (Preliminary to Clinical Trial). Demonstrate usability with iterative user assessment testing in a clinical setting.

Specific Aim 3. Test the clinical efficacy of VidaTalk via android application with MV patients by examining qualitative and quantitative endpoints in a clinical setting. Aim 3 hypothesis: MV patients using VidaTalk will demonstrate notable reductions in patient-reported frustration and communication difficulty, anxiety, sedation exposure, delirium/coma-free days, and improved patient and family satisfaction with ICU care compared to MV patients receiving attention-control.

Specific Aim 4. Validation of electronic visual analogue scale, versus current standard paper scale.

Specific Aim 5. Test the effect of the communication tablet (VidaTalk) on psychological symptoms in family caregivers.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

1. ≥18 years old
2. Able to communicate in English
3. Awake alert, responding appropriately to commands.
4. Normal (aided or unaided) hearing and vision
5. Able to control head, arm and hand movements
6. Physiologically stable and in no acute distress (per nurse report)

Exclusion Criteria:

1. Pre-existing communication impairments
2. Diagnosis of severe dementia or brain injury
3. CAM-ICU positive for delirium
4. unresponsiveness or inattention

Aim 2:

Inclusion Criteria:

1. ≥18 years old
2. Able to communicate in English
3. Awake alert, responding appropriately to commands.
4. Normal (aided or unaided) hearing and vision
5. Able to control head, arm and hand movements
6. Physiologically stable and in no acute distress (per nurse report)
7. Intubated via oral endotracheal or tracheal tube without speaking valve, receiving mechanical ventilation

Exclusion Criteria:

1. Pre-existing communication impairments
2. Diagnosis of severe dementia or brain injury
3. CAM-ICU positive for delirium
4. unresponsiveness or inattention

Aim 3:

Inclusion Criteria:

1. ≥18 years old
2. Able to communicate in English
3. Awake alert, responding appropriately to commands.
4. Normal (aided or unaided) hearing and vision
5. Able to control head, arm and hand movements
6. Physiologically stable and in no acute distress (per nurse report)
7. Intubated via oral endotracheal or tracheal tube without speaking valve, received mechanical ventilation during past 48 hours

Exclusion Criteria:

1. Pre-existing communication impairments
2. Diagnosis of severe dementia or brain injury
3. CAM-ICU positive for delirium
4. unresponsiveness or inattention

Aim 5

Inclusion Criteria:

1. Family caregivers of patient participants enrolled in Aim 3 as identified by the patient or self
2. >/=18 years old
3. Able to read and speak English
4. Non-professional, unpaid caregiver
5. Plans to visit at least 3 days/ week during ICU stay
6. Reliable telephone access (for follow-up assessment)

Exclusion Criteria:

1. Age under 18 years
2. Unable to read and speak English
3. Severe uncorrected hearing loss
4. Self-reported diagnosis of dementia or Alzheimer's
5. Self-reported psychiatric disorder (bipolar disorder, schizophrenia) or substance abuse requiring inpatient treatment within the last 12 months
6. Unreliable telephone access

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Happ, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility by critical care research coordinators and referred to the study coordinator and research assistant for bedside eligibility screening and recruitment.
Groups:
- Aim 1- VidaTalk Post-extubation: Aim 1 is a two group iterative design preliminary to clinical trial. Group 1 & 2 will each consist of five previously mechanically ventilated patients who will be recruited from the ICUs at the OSUMC including discharged patients.
  Group 1 will use an initial android prototype of VidaTalk tablet application to be assessed for functionality (ergonomics, ease of use, ease of learning, simplicity, effectiveness and user interface) and usability on customizable communication, picture symbols, and integration with mobile communication devices.
  Group 2 will use an improved alpha prototype of VidaTalk tablet application version engineered from observations made during Group 1 sessions.
  Aim 1 - VidaTalk - post-extubation: Observation of task completion will be made while patients complete a series of messages using the VidaTalk app:
  * Tell me you are tired
  * Tell me you are having pain
  * Rate this pain
  * Tell me there is pain in your back
  * Tell me your pain is sharp
  * Ask to see
- Aim 2 - VidaTalk Intubated: Usability testing preliminary to Clinical Trial. Mechanically Ventilated patients will provide feedback on acceptability, will perform test messages with minimal errors, and will rate VidaTalk an overall average score of 4.5 or higher (Likert-type scale; 1 to 7) on usability questions. Prior to implementing these procedures, the company will perform further iterative design assessments and engineer a Vidatalk tablet application prototype. This prototype will be used with a final group of ten (10) intubated patients receiving mechanical ventilation support to field-test the prototype for functionality (human-device interaction factors, feasibility, and usability) and acceptability.
  Intervention is usability tasks with the VidaTalk app
  Aim 2 - VidaTalk - intubated: Usability testing prior to clinical trial. The company will have performed further iterative design assessments and engineered a Vidatalk tablet application prototype for a field-test for functionality (human-
- Nurse Focus Group - PreClinical Trial Phase: ICU nurses were recruited to participate in qualitative focus group interviews regarding their impressions of the VidaTalk tablet app for use with mechanically ventilated patients, their experience (if any) of using the app, and general perspectives about communicating with mechanically ventilated ICU patients. We also elicited suggestions for app improvement. Group interviews were conducted by the PI in a hospital conference room away from patient care.
- Aim 3 - VidaTalk Tablet App: Test the clinical efficacy of VidaTalk with MV patients by examining qualitative & quantitative endpoints in a clinical setting. 35 intubated patients (oral endotracheal tube or tracheostomy) will be randomized to the intervention arm and will receive a protocolized instruction in the use of the VidaTalk application including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 minutes) each day to check user needs and concerns and will review or retrain on message options if needed.
  Intervention will be receipt of VidaTalk tablet application.
  Aim 3 - VidaTalk tablet app: Patients in the intervention group will receive a protocolized instruction in the use of the VidaTalk application and mounting of the device including patient return demonstration.
- Aim 3 - Attention-control: 35 intubated patients (oral endotracheal tube or tracheostomy) will receive the standard of care, which may include primarily writing tools (paper and pen) and, occasionally, picture or alphabet communication charts.
  Patients randomized to the control group will receive a protocolized introduction to the bedside Android device without the VidaTalk application, focusing instead on a common tablet application. Daily visits will be conducted with control group patients to query on use of the attention-control tablet.
  Interventions will be Aim 3 - attention-control with non-VidaTalk tablet.
  Aim 3 - attention-control with non-VidaTalk tablet: Patents randomized to the control group will receive a protocolized introduction to the bedside Android device without the VidaTalk app, focusing instead on a common tablet application. Daily visits will be conducted with control group patients to query on use of the attention-control tablet.
- Nurse Focus Group - VidaTalk RCT: ICU Nurses who had experience with using the VidaTalk tablet app with mechanically ventilated patients were recruited to participate in focus group interviews to obtain their perspectives and experience on using the application as well as suggestions for app improvement. Group interviews were conducted by the PI in a hospital conference room away from patient care.
- Aim 5-VidaTalk Efficacy in Family Caregivers - VidaTalk Group: Aim 5 will test the preliminary efficacy of VidaTalk compared to attention control (AC) on anxiety and depression symptoms in family caregivers during the ICU stay and post-discharge (1-mos; 3-mos; 6-mos) and PTSD-related symptoms post-discharge both qualitatively and quantitatively.
  Aim 5.a.) Psychological outcomes (anxiety, depression, and PTSD-related symptoms) between the two groups will be compared at each time point and across time. Aim 5.b.) Family caregivers' perceived communication difficulty will be measured .Aim 5.c.) Family caregivers' experience of communication while they were visiting the patient who received the VidaTalk app in the ICU and their emotional reactions to communication with a patient will be measured.
  VidaTalk (Intervention) Group receives brief introduction, instruction sheet and completes ICU bedside visitation log with dates and times of visits.
- Aim 5 Family Caregiver - Attention Control: Usual care condition for family communication with mechanically ventilated patients. Family caregivers receive tablet instruction sheet (no VidaTalk app). Family caregivers were asked to enter dates and times of visits into ICU bedside visitation log.
Period: Overall Study
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Nurse Focus Group - PreClinical Trial Phase | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Nurse Focus Group - VidaTalk RCT | Aim 5-VidaTalk Efficacy in Family Caregivers - VidaTalk Group | Aim 5 Family Caregiver - Attention Control
Started | 13 | 23 | 7 | 31 | 32 | 7 | 18 | 16
Completed | 11 | 15 | 7 | 23 (Completed Primary outcome (daily measures) = 27 Completed Secondary outcomes (@ICU discharge) = 23) | 26 (Completed Primary outcome (daily measures) = 27 Completed Secondary outcomes (@ICU discharge) = 26) | 5 | 7 (At discharge/ extubation =11 1-mos post-discharge = 8 3-mos post-discharge = 8) | 9 (At discharge/ extubation =15 1-mos post-discharge = 12 3-mos post-discharge = 11)
Not Completed | 2 | 8 | 0 | 8 | 6 | 2 | 11 | 7
Not completed — patient deterioration, fatigue | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 1 | 0 | 8 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — extubation or early discharge | 0 | 0 | 0 | 5 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 6

BASELINE CHARACTERISTICS:
Population: missing data on two patients in Aim 1 who dropped out
Groups:
- Aim 1- VidaTalk Post-extubation: Preliminary to clinical trial. Grp1+ Grp2 will each consist of five previously mechanically ventilated patients recruited from the ICUs at the OSUWMC.
  Grp 1 will use an initial android prototype of VidaTalk tablet application assessed for functionality + usability on a series of scripted communication tasks.
  Grp 2 will use an improved alpha prototype of VidaTalk tablet application version engineered from observations made during Grp 1 sessions.
  Aim 1 - VidaTalk - post-extubation: Observation of task completion will be made while patients complete messages using the VidaTalk app:
  Tired, Pain - rating, location, quality, Ask for doctor, Finger writing, Keyboard phrase. Patients will also complete 1-item difficulty rating + 3-item After-Scenario Questionnaire after each task.
  Patients will rate the extent to which they would use the device if they were an ICU patient unable to speak.
  Grp 1 only: will be asked their preferences for customizing the app.
- Aim 5-VidaTalk Efficacy in Family Caregivers- VidaTalk Group: Aim 5 will test the preliminary efficacy of VidaTalk compared to attention control (AC) on anxiety and depression symptoms in family caregivers during the ICU stay and post-discharge (1-mos; 3-mos; 6-mos) and PTSD-related symptoms post-discharge both qualitatively and quantitatively.
  Aim 5.a.) Psychological outcomes (anxiety, depression, and PTSD-related symptoms) between the two groups will be compared at each time point and across time. Aim 5.b.) Family caregivers' perceived communication difficulty will be measured Aim 5.c.) Family caregivers' experience of communication while they were visiting the patient who received the VidaTalk app in the ICU and their emotional reactions to communication with a patient will be measured.
- Aim 5 Family Caregiver- Attention Control: Usual care condition for family communication with mechanically ventilated patients. Family caregivers receive tablet instruction sheet (no VidaTalk app). Family caregivers were asked to enter dates and times of visits into ICU bedside visitation log.
- Total: Total of all reporting groups
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers- VidaTalk Group | Aim 5 Family Caregiver- Attention Control | Total
Number analyzed (Participants) | 13 | 23 | 31 | 32 | 18 | 16 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is measured in years, information collected from electronic medical record for patient age. Family age was self-reported.
  Cumulative age average is calculated for Aim 3 RCT only, n=63 ICU patients. Not on 133 participants. Family participants and pre-RCT patient data are removed.
  years | 55.92 (15.4) | 57.57 (13.41) | 52.1 (13.7) | 53.6 (14.7) | 48.94 (15.84) | 50.69 (15.89) | 52.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — categorical male, female. Patient data from electronic medical record. Family caregiver self-report.
  Participants
    Female | 5 | 9 | 13 | 12 | 15 | 15 | 69
    Male | 8 | 14 | 18 | 20 | 3 | 1 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — NIH ethnicity categories
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 13 | 23 | 31 | 32 | 18 | 16 | 133
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — NIH Categories applied
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 5 | 4 | 5 | 3 | 19
    White | 12 | 20 | 26 | 28 | 12 | 13 | 111
    More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants] — dichotomized high school graduate or less; some college Population: number analyzed differs from overall due to missing data
  Participants
    number analyzed (Participants) | 11 | 19 | 31 | 32 | 18 | 16 | 127
    High school graduate or less | 4 | 12 | 19 | 13 | 5 | 5 | 58
    Some college | 7 | 7 | 12 | 19 | 13 | 11 | 69
severity of illness [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology, Age, and Chronic Health Evaluation (APACHE) iii severity of illness scale for critical illness - age, acute physiology and chronic illness weighted scores. Scores range from 0 to 299, with larger scores indicating more severe illness and higher risk of death. Weighted subscales for acute physiology, age and chronic health are summed to determine total score. Population: not applicable to this arm
  Total analysis is limited to RCT Aim 3, n=63 patients. Pre-RCT data removed as not applicable.
  units on a scale
    number analyzed (Participants) | 11 | 15 | 31 | 32 | 0 | 0 | 89
    (all) | 65.0 (17.82) | 72.8 (26.55) | 75.6 (21.8) | 77.0 (27.2) |  |  | 76.3 (24.5)
Intubation Method [Count of Participants; unit: Participants] — Dichotomous - oral intubation or tracheostomy Population: not applicable to extubated patients and family caregiver arm
  Participants
    number analyzed (Participants) | 0 | 19 | 31 | 32 | 0 | 0 | 82
    oral intubation |  | 8 | 15 | 16 |  |  | 39
    tracheostomy |  | 11 | 16 | 16 |  |  | 43
Physical Restraint [Count of Participants; unit: Participants] — dichotomous yes (presence of wrist restraint) vs. no restraint Population: Only measured for patients in the RCT, Aim 3
  Participants
    number analyzed (Participants) | 0 | 0 | 31 | 32 | 0 | 0 | 63
    (all) |  |  | 5 | 8 |  |  | 13
Patient Anxiety [Mean (Standard Deviation); unit: units on a scale] — Visual Analogue scale (VAS) anxiety 0-10 scale was used on Aim 3 only. Self report of anxiety using Visual Analog Scale-Anxiety (VAS-A) 0-10 scale on a 100-mm scale was used to measure anxiety. Higher scores indicate greater severity of anxiety. 100 mm scale was divided by 10 to reach the 0-10 scale. Population: not assessed in preclinical group
  units on a scale
    number analyzed (Participants) | 0 | 0 | 31 | 32 | 0 | 0 | 63
    (all) |  |  | 5.9 (3) | 6.4 (3.1) |  |  | 6.2 (3.0)
Patient Communication Difficulty [Mean (Standard Deviation); unit: units on a scale] — Single item rating, patient self-report 0= not at all to 4= extremely difficult Population: Patient measure only. Not applicable in Aim 5
  Total mean calculation limited to RCT Aim 3 only, n=63 patients. Pre-RCT data removed as not applicable
  units on a scale
    number analyzed (Participants) | 11 | 18 | 31 | 32 | 0 | 0 | 92
    (all) | 3.8 (0.63) | 3.33 (0.84) | 3.1 (1.2) | 3.4 (0.9) |  |  | 3.3 (1.1)
Patient Frustration with Communication [Mean (Standard Deviation); unit: units on a scale] — single item rating scale, patient self-report. 0= not at all to 4 = extremely frustrating Population: Data missing on dropouts in Aim 1 and 2. Patient measure only, not applicable to Aim 5
  Total mean calculation limited to RCT Aim 3 only, n=63 patients. Pre-RCT data removed as not applicable
  units on a scale
    number analyzed (Participants) | 11 | 18 | 31 | 32 | 0 | 0 | 92
    (all) | 3.6 (1.26) | 2.94 (1.35) | 3.4 (1.0) | 3.9 (0.3) |  |  | 3.6 (0.7)
Family Caregiver Anxiety [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) Anxiety sub scale including 7 items each scored from 0-3 with total scores ranging from 0 - 21 with higher scores indicating higher levels of anxiety. Population: not assessed in patient samples, only Aim 5
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 16 | 34
    (all) |  |  |  |  | 9.22 (5.02) | 9.25 (4.49) | 9.24 (4.71)
Family Caregiver Depression [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS-D)- Depression Subscale including 7 items each scored from 0-3 with total scores ranging from 0 - 21 with higher scores indicating higher levels of depression symptoms. Population: HADS not assessed in patient samples, only Aim 5
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 16 | 34
    (all) |  |  |  |  | 5.89 (3.85) | 5.25 (4.17) | 5.59 (3.96)
Family Communication Survey [Mean (Standard Deviation); unit: units on a scale] — Family Communication Survey is an investigator developed measure. Self-report measure of perceived difficulty communicating with mechanically ventilated patients. This tool contains nine items, and each item is scored on a five-point Likert scale (1, strongly disagree; 2, disagree; 3, not sure; 4, agree; and 5, strongly agree). Total scores range from 9 to 45, and higher scores indicate less perceived communication difficulty. Item 9 score was reversed for a total score. Population: Measure is for Family caregivers only, Aim 5
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 16 | 34
    (all) |  |  |  |  | 25.94 (6.24) | 24.93 (5.57) | 25.47 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Patient-reported Communication Difficulty Rating Using Single Item 0-4 Rating Scale
Description: Aim 3 - Mean item score of daily by patient self report using a single item Likert-type scale from the Ease of Communication Scale (ECS) where scores range from 0 "not hard at all" to 4 "extremely hard"
Time Frame: Daily post-randomization until extubation or ICU discharge up to maximum of 28 days in the ICU
Population: This outcome is only for the clinical trial. Applies only to Aim 3 arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aim 2 - VidaTalk Intubated: Usability testing preliminary to Clinical Trial (Aim 3). Mechanically Ventilated patients will provide feedback on acceptability, will perform test messages with minimal errors, and will rate VidaTalk an overall average score of 4.5 or higher (Likert-type scale; 1 to 7) on usability questions. Prior to implementing these procedures, the company will perform further iterative design assessments and engineer a Vidatalk tablet application prototype. This prototype will be used with a final group of ten intubated patients receiving mechanical ventilation support to field-test the prototype for functionality (human-device interaction factors, feasibility, and usability) and acceptability.
  Intervention is usability tasks with the VidaTalk app
  Aim 2 - VidaTalk - intubated: Usability testing prior to clinical trial. The company will have performed further iterative design assessments and engineered a Vidatalk tablet application prototype for a field-test for functionality (human-
- Aim 3 - VidaTalk Tablet App: Test the clinical efficacy of VidaTalk with MV patients by examining qualitative and quantitative endpoints in a clinical setting. 35 intubated patients (oral endotracheal tube or tracheostomy) will be randomized to the intervention arm and will receive a protocolized instruction in the use of the VidaTalk application including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 min) each day to check user needs and concerns and will review or retrain on message options if needed.
  Intervention will be receipt of VidaTalk tablet application.
  Aim 3 - VidaTalk tablet app: Patients in the intervention group will receive a protocolized instruction in the use of the VidaTalk application and mounting of the device including patient return demonstration.
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 25 | 25 | 0
score on a scale |  |  | 3.10 (1.98) | 3.28 (1.90) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = .18

2. Secondary Outcome: Mean Patient Reported Anxiety Score Using Visual Analogue Scale
Description: Aim 3 - Calculated mean of daily measure by patient mark (x) or point on the Visual Analogue Scale for anxiety, a 100 mm vertical line ranging from 0 ("not anxious at all") to 10 ("most anxious I've ever been").
Time Frame: Daily post-randomization until extubation or ICU discharge up to maximum of 28 days in the ICU
Population: This Secondary Outcome is for participants in Aim 3 only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aim 1- VidaTalk Post-extubation: Aim 1 - two group iterative design preliminary to clinical trial. Group 1/Group 2 will each consist of five previously mechanically ventilated patients who will be recruited from the ICU at the Ohio State University including discharged patients. Group 1 will use an android prototype of VidaTalk tablet application to be assessed for functionality (ergonomics, ease of use, ease of learning, simplicity, effectiveness and user interface) and usability on customizable communication, picture symbols, and integration with mobile communication devices.Group 2 will use an improved alpha prototype of VidaTalk tablet application version engineered from observations made during Group 1 sessions. Aim 1 - VidaTalk - post-extubation: Observation of task completion will be made while patients complete a series of messages using the VidaTalk app:Tell me you are tired; Tell me you are having pain; Rate this pain; Tell me there is pain in your back; Tell me your pain is sharp; Ask to see the doctor; Write your favorite color by drawing with your finger; Type "How are you?"
  Patients will also complete a 1-item difficulty rating and a 3-item After-Scenario Questionnaire (ASQ) after each task. Patients will also be asked to a) comment on the customization of the app and make suggestions; b) rate the extent to which they would use the device if they were an ICU patient and unable to speak. Group 1 only:
  Patients will be asked about their preferences for customizing the VidaTalk app.
- Aim 2 - VidaTalk Intubated: Usability testing preliminary to Clinical Trial (Aim 3). Mechanically Ventilated patients will provide feedback on acceptability, will perform test messages with minimal errors, and will rate VidaTalk an overall average score of 4.5 or higher (Likert-type scale; 1 to 7) on usability questions. Prior to implementing these procedures, the company will perform further iterative design assessments and engineer a Vidatalk tablet application prototype. This prototype will be used with a final group of ten (10) intubated patients receiving mechanical ventilation support to field-test the prototype for functionality (human-device interaction factors, feasibility, and usability) and acceptability.
  Intervention is usability tasks with the VidaTalk app
  Aim 2 - VidaTalk - intubated: Usability testing prior to clinical trial. The company will have performed further iterative design assessments and engineered a Vidatalk tablet application prototype for a field-test for functionality (human-device interaction factors, feasibility, and usability) and acceptability. Data will be collected by a trained data collector as in Aim 1 with the addition of Ease of Communication and Frustration ratings before and after the testing sequence. To reduce burden, patients in this group will complete the 3-item ASQ one time after all tasks are completed. They will also complete a 13-item System Usability Scale (SUS).
- Aim 3 - VidaTalk Tablet App: Test the clinical efficacy of VidaTalk with MV patients by examining qualitative and quantitative endpoints in a clinical setting. 35 intubated patients (oral endotracheal tube or tracheostomy) will be randomized to the intervention arm and will receive a protocolized instruction in the use of the VidaTalk application including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 minutes) each day to check user needs and concerns and will review or retrain on message options if needed.
  Intervention will be receipt of VidaTalk tablet application.
  Aim 3 - VidaTalk tablet app: Patients in the intervention group will receive a protocolized instruction in the use of the VidaTalk application and mounting of the device including patient return demonstration of key features, and review/ testing to competence conducted by a trained interventionist. When available, a family member may be included in surveys about the patients hospital stay, if patient agrees. The interventionist will visit patients briefly (5-10 minutes) each day to check user needs and concerns and will review or retrain on message options if needed.
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 25 | 25 | 0
score on a scale |  |  | 5.55 (6.54) | 6.02 (6.07) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = .48

3. Secondary Outcome: Mean Patient Frustration With Communication
Description: Aim 3 - This will be the calculated mean of the daily Communication Frustration scale - a single item scale reported by the patient, ranging from 0 "not frustrating" to 4 "extremely frustrating"
Time Frame: Daily post-randomization until extubation or ICU discharge up to maximum of 28 days in the ICU
Population: This information is for Aim 3 only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 25 | 25 | 0
units on a scale |  |  | 3.14 (1.89) | 3.53 (0.17) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Other; p = 0.10, Effect size; Effect size =-0.29
Statistical Analysis 2: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = .10, t-test, 2 sided; Mean Difference (Final Values) = 0.39

4. Secondary Outcome: Mean Daily Sedation Exposure
Description: Used in Aim 3 only. Calculation of benzodiazepine and morphine equivalents (for opiates) using hospital conversion charts (pharmacy conversion chart). All benzo IV doses were converted to Lorazepam IV doses. All opioid IV doses were converted to morphine IV doses. All benzo oral doses were converted to Lorazepam oral doses. All opioid oral doses were converted to morphine oral doses. Oral doses were converted to IV equivalents. Summed doses of Lorazepam IV and morphine IV were calculated for each study day for each patient. Doses were converted to milligrams per kilogram based on the patient's body weight. Higher numbers indicate greater sedation and/or opiate exposure.
Time Frame: Daily post-randomization until extubation or ICU discharge up to maximum of 28 days in the ICU daily in ICU
Population: P-values were derived from mixed-effects regression using rank-based sedation exposure
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 29 | 27 | 0
mg/kg
  Benzo (mg/kg) |  |  | .01 (.05) | .008 (.02) |
  Morphine (mg/kg) |  |  | .84 (2.10) | .24 (.50) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Benzodiazepine exposure; Test type: Superiority; p = 0.02, Mixed Models Analysis
Statistical Analysis 2: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Opioid Exposure; Test type: Superiority; p = 0.291, Mixed Models Analysis

5. Secondary Outcome: Ease of Communication at Extubation /ICU Discharge
Description: Ease of Communication Scale -10-item likert scale total score ranging from 0-40. Each item is 0-4 likert scale, total score is sum of all items with higher scores indicating greater communication difficulty.
Time Frame: measured at Extubation /ICU Discharge
Population: Extubated ICU patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 16 | 26 | 0
score on a scale |  |  | 23.19 (11.31) | 27.23 (10.46) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.38, t-test, 2 sided; Mean Difference (Final Values) = 3.04

6. Secondary Outcome: Percentage of Patients Scoring in the "Calm" Range During Study Days on Richmond Agitation Sedation Score
Description: The Richmond Agitation Sedation Scale, a 10-level observational rating of agitation-sedation motor activity ranging from +4 'combative' to -5 unresponsive, with 0 as calm. Since this is a categorical measure, we compared proportion of patients with RASS in -1 to +1 (calm) range during study days.
Time Frame: Daily post-randomization until extubation or ICU discharge up to maximum of 28 days in the ICU
Population: Since this is a categorical measure, we compared percentage of patients with RASS in -1 to +1 (calm) range during study days.
Measure: Number; unit: percentage of participants in calm range
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 27 | 27 | 0
percentage of participants in calm range |  |  | 81.48 | 77.78 |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.32, Chi-squared

7. Secondary Outcome: Delirium/Coma -Free Days
Description: Aim 3 -Delirium/coma-free days is defined as the number of days alive and free of delirium and coma during the 28-day study period. Delirium will be coded as present when a patient displays both features 1 and 2, and either 3 or 4 of the CAM-ICU (Confusion Assessment Method). Coma is defined as a RASS (Richmond Agitation-Sedation Scale ) assessment score of -4 or -5.
Time Frame: Daily, from enrollment to 28 days post-enrollment
Population: Calculated as % days with delirium/total ICU days.
Measure: Number; unit: percent days with delirium/total ICU day
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 27 | 27 | 0
percent days with delirium/total ICU day |  |  | 8.26 | 8.54 |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.93, Mixed Models Analysis; Odds Ratio (OR) = .93, 95% CI 2-sided [0.19 to 4.72]

8. Secondary Outcome: Family Satisfaction With Care in the Intensive Care Unit FS-ICU
Description: (Aim3 )The Family Satisfaction with ICU Care (FS-ICU 24R) questionnaire overall satisfaction score is derived from questions 1 through 24 (26 items) and combines two subscale summary scores. The satisfaction with care summary score is derived from the questions numbered 1 through 14 (which consists of 16 questions because question 2 has parts a, b and c). The satisfaction with decision making summary score is derived from questions 15 through 24 (10 questions). All questions are coded as integers from 1 (worst) to 5 (best). Rescale the summary scores from 1 through 5 to 0 through 100 by subtracting 1 from the scores (so they can range from 0 to 4) and then multiplying each score by 25.
Time Frame: One 10 minute survey will be given at patient's ICU discharge or extubation
Population: Total score on the Family Satisfaction in the Intensive Care Unit Survey (FS-ICU) completed by designated family caregiver-support person.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 8 | 8 | 0
score on a scale |  |  | 81.8 (13.8) | 92.4 (7.2) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = 10.6

9. Secondary Outcome: Electronic Visual Analogue Scale-validation Measure
Description: (Aim4) visual analogue touch screen scale via android tablet with REDCap link.
  Not able to calculate because the touch screen scale was unreliable. Patients often needed assistance with the touch screen cursor for this experimental measure. We determined that pencil and paper analogue scale was superior for this patient population.
Time Frame: Only measured at baseline, order of administration randomized before or after paper version
Population: Not able to calculate because the touch screen scale was unreliable. Patients often needed assistance with the touch screen cursor for this experimental measure. We determined that pencil and paper analogue scale was superior for this patient population.
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Patient Satisfaction With Care
Description: A 24-item survey with lower scores indicating greater satisfaction with care.
Time Frame: Measured at extubation or discharge from ICU which ever comes first
Population: Patient Satisfaction with Care at extubation /ICU discharge single item likert type scale 1 (very dissatisfied) to 5 (very satisfied)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 22 | 25 | 0
units on a scale |  |  | 4.45 (1.01) | 4.56 (0.92) |
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.71, t-test, 2 sided

11. Secondary Outcome: Family Member Anxiety
Description: (Aim 5) Hospital Anxiety and Depression Scale (HADS) Anxiety sub scale including 7 items each scored from 0-3 with total scores ranging from 0 - 21 with higher scores indicating higher levels of anxiety.
Time Frame: Baseline, patient extubation or discharge from ICU, 1-month, 3-month, 6-month post-discharge
Population: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aim 5-VidaTalk Intervention for Family Members: Aim 5 - Vida Talk Intervention with Family Members
- Aim-5 Control Group: Aim - 5 Control Group
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Intervention for Family Members | Aim-5 Control Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 14
units on a scale
  Baseline |  |  |  |  | 9.14 (5.08) | 9.29 (4.83)
  Patient Extubation or Discharge from ICU: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 13
  Patient Extubation or Discharge from ICU |  |  |  |  | 8.67 (4.44) | 9.62 (4.86)
  1-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 12
  1-month |  |  |  |  | 4.86 (4.06) | 9.17 (4.80)
  3-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 10
  3-month |  |  |  |  | 6.83 (4.92) | 6.80 (5.07)
  6-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 9
  6-month |  |  |  |  | 6.80 (5.63) | 6.22 (6.48)
Statistical Analysis 1: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; Baseline; Test type: Superiority; p = 0.94, t-test, 2 sided
Statistical Analysis 2: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; Patient Extubation or Discharge from ICU; Test type: Superiority; p = 0.89, t-test, 2 sided
Statistical Analysis 3: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; 1-Month; Test type: Superiority; p = 0.38, t-test, 2 sided
Statistical Analysis 4: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; 3-Month; Test type: Superiority; p = 0.63, t-test, 2 sided
Statistical Analysis 5: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; Test type: Superiority; p = .73, t-test, 2 sided

12. Secondary Outcome: Family Member Depression
Description: (Aim 5). Hospital Anxiety and Depression Scale (HADS-D)- Depression Subscale including 7 items each scored from 0-3 with total scores ranging from 0 - 21 with higher scores indicating higher levels of depression symptoms.
Time Frame: Baseline, patient extubation or discharge from ICU, 1-month, 3-month, 6-month post-discharge
Population: Aim 5 Family member depression HADS-D subscale
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aim 5-VidaTalk Intervention for Family Members: Aim 5 - VidaTalk Intervention for Family Members
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Intervention for Family Members | Aim-5 Control Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 14
units on a scale
  Baseline |  |  |  |  | 5.86 (3.98) | 5.50 (4.31)
  Patient Extubation or Discharge from ICU: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 13
  Patient Extubation or Discharge from ICU |  |  |  |  | 5.78 (4.32) | 5.15 (4.43)
  1-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 12
  1-month |  |  |  |  | 7.43 (2.64) | 6.20 (3.73)
  3-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 10
  3-month |  |  |  |  | 7.03 (3.98) | 5.53 (3.93)
  6-month: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 9
  6-month |  |  |  |  | 6.33 (4.27) | 4.33 (3.67)
Statistical Analysis 1: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; Baseline; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 2: Comparison: Aim 5-VidaTalk Intervention for Family Members; Patient extubation or discharge from ICU; Test type: Superiority; p = 0.84, t-test, 2 sided
Statistical Analysis 3: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; 1-month; Test type: Superiority; p = 0.96, t-test, 2 sided
Statistical Analysis 4: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; 3-Month; Test type: Superiority; p = 0.17, t-test, 2 sided
Statistical Analysis 5: Comparison: Aim 5-VidaTalk Intervention for Family Members vs Aim-5 Control Group; Test type: Superiority; p = .39, t-test, 2 sided

13. Secondary Outcome: Post-traumatic Stress Symptoms: Impact of Events Scale-revised (IES-R)
Description: (Aim 5) Impact of Events Scale-revised. The IES-R is a 22-item self-report instrument with three subscales including intrusion (8 items), avoidance (8 items), and hyperarousal (6 items). The respondent is asked to report the degree of distress experienced for each item in the past 7 days. Each item is scored on a five-point Likert scale (0, not at all; 1, rarely; 2, occasionally; 3, fairly often; and 4, often) and total scores range from 0 to 88. Higher scores are representative of greater distress.
Time Frame: 1-month, 3-month, 6-month post-discharge
Population: Impact of events scale median/IQR
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Aim-5 Control Group: Aim 5 - Control Group
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers | Aim-5 Control Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 12
units on a scale
  1-month |  |  |  |  | 21.5 [1.5 to 33.5] | 30.5 [11 to 48]
  3-months: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 10
  3-months |  |  |  |  | 21 [4.75 to 31.00] | 27.5 [18 to 41.25]
  6-months: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 9
  6-months |  |  |  |  | 23 [15.50 to 37.50] | 26 [15 to 49]
Statistical Analysis 1: Comparison: Aim 5-VidaTalk Efficacy in Family Caregivers vs Aim-5 Control Group; 1-month; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Aim 5-VidaTalk Efficacy in Family Caregivers vs Aim-5 Control Group; 3-month; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Aim 5-VidaTalk Efficacy in Family Caregivers vs Aim-5 Control Group; 6-month; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Family Communication Difficulty
Description: Family Communication Survey administered to participant families. Sum of 9-items with each item rating 0 (not at all) to 4 (extremely difficult), resulting in a total summed score from 0 - 36. Higher scores indicate greater difficulty.
Time Frame: baseline and extubation or discharge from the ICU
Population: Family Communication Survey baseline and extubation or discharge from the ICU
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aim 5-VidaTalk Intervention in Family Members: Aim 5 - VidaTalk Intervention in family members
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Intervention in Family Members | Aim-5 Control Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 14
units on a scale
  Baseline |  |  |  |  | 28.67 (2.27) | 25.62 (1.59)
  Extubation or Discharge from ICU: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 13
  Extubation or Discharge from ICU |  |  |  |  | 33.67 (1.60) | 29.46 (1.20)

15. Secondary Outcome: Communication Task Error Rate
Description: Aims 1 & 2 - count of the number of errors recorded by video screen capture for each of 8 communication tasks. Individual patients ranged from 0 to 9 errors, however this measure contains no upper range per task as it is a count of actual observed errors committed by patients.
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion. This outcome applies only to Aim 1 & 2 arms.
Population: Aim 1 extubated patients. Using group 1 and group 2 summary data, 11 patients completed 82 tasks (6 were abandoned, 5 of these by one patient). Removing abandonments.
Measure: Number; unit: Errors
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 11 | 11 | 0 | 0 | 0
Errors
  Task 1 (Tired) | .45 | 1.09 |  |  |
  Task 2 (Pain) | .09 | 1.0 |  |  |
  Task 3 (Pain Rating) | .273 | 1.0 |  |  |
  Task 4 (Pain Location ): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 4 (Pain Location ) | .30 | .36 |  |  |
  Task 5 (Pain Quality): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 5 (Pain Quality) | .40 | .63 |  |  |
  Task 6 (Doctor): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 6 (Doctor) | .20 | 1.18 |  |  |
  Task 7 (Word Draw): number analyzed (Participants) | 9 | 11 | 0 | 0 | 0
  Task 7 (Word Draw) | .22 | .18 |  |  |
  Task 8 (Typing): number analyzed (Participants) | 10 | 10 | 0 | 0 | 0
  Task 8 (Typing) | .50 | .50 |  |  |

16. Secondary Outcome: Total Error Rate
Description: Aims 1 & 2 - calculated mean of the total number of errors recorded by video screen capture divided by the number of communication tasks completed (8 maximum) Aim 1 extubated patients. Using group 1 and group 2 summary data, 11 patients completed 82 tasks (6 were abandoned, 5 of these by one patient). Removing abandonments, total number of errors = 25/ 82 tasks = 0.30 error rate.
  Aim 2 intubated patients. 11 patients completed 69 tasks (18 were abandoned; 1 task was refused). Removing abandonments, total number of errors = 60/ 69 tasks = 0.87error rate.
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion
Population: Aim 1 extubated patients. Using group 1 and group 2 summary data, 11 patients completed 82 tasks (6 were abandoned, 5 of these by one patient).
  Aim 2 intubated patients. 11 patients completed 69 tasks (18 were abandoned; 1 task was refused).
Measure: Number; unit: error rate
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 11 | 11 | 0 | 0 | 0
error rate | 0.30 | 0.87 |  |  |

17. Secondary Outcome: Patient Satisfaction With Communication Task Ease
Description: Aims 1 & 2 - a single item from the After Scenario Questionnaire (ASQ) of patient's self rating of satisfaction with the "ease of completing" each of 8 communication tasks on the usability test. Question asked of patients was "Overall, I am satisfied with the ease of completing this task". 1-strongly disagree 7-strongly agree. Higher scores indicated greater satisfaction with the ease of completing the task.
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion
Population: Aim 1 Extubated patients - mean Task Ease Rating Aim 2 Intubated patients - mean Task Ease Rating
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 11 | 11 | 0 | 0 | 0
score on a scale
  Task 1 (Tired): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 1 (Tired) | 5.7 (1.85) |  |  |  |
  Task 2 (Pain): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 2 (Pain) | 6.7 (0.647) |  |  |  |
  Task 3 (Pain Rating): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 3 (Pain Rating) | 6.7 (0.675) |  |  |  |
  Task 4 (Pain Location): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 4 (Pain Location) | 6.7 (0.675) |  |  |  |
  Task 5 (Pain Quality): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 5 (Pain Quality) | 6.9 (0.316) |  |  |  |
  Task 6 (Doctor): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 6 (Doctor) | 5.8 (1.68) |  |  |  |
  Task 7 (Draw Word): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 7 (Draw Word) | 6.9 (0.316) |  |  |  |
  Task 8 (Typing): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 8 (Typing) | 5.9 (2.08) |  |  |  |
  Overall Ease: number analyzed (Participants) | 0 | 11 | 0 | 0 | 0
  Overall Ease |  | 5.82 (1.60) |  |  |

18. Secondary Outcome: Observed Task Completion Time (in Seconds)
Description: Aims 1 & 2 - This is the time, measured in seconds, on the screen capture recording beginning with the communication task command to patient completion of the communication task or message to patient completion of each of the 8 communication tasks on the usability test, calculated from the screen capture recordings
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion
Population: This is the time, measured in seconds, on the screen capture recording beginning with the communication task command to patient completion of the communication task or message to patient completion of each of the 8 communication tasks on the usability test, calculated from the screen capture recordings
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 11 | 11 | 0 | 0 | 0
seconds
  Task 1 (Tired) | 64.27 (69.02) | 117.45 (107.29) |  |  |
  Task 2 (Pain) | 16.73 (13.06) | 80.0 (143.62) |  |  |
  Task 3 (Pain Rating): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 3 (Pain Rating) | 26.6 (26.71) | 74.0 (64.35) |  |  |
  Task 4 (Pain Location): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 4 (Pain Location) | 25.3 (34.19) | 34.82 (34.19) |  |  |
  Task 5 (Pain Quality): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 5 (Pain Quality) | 44.0 (75.83) | 52.73 (49.26) |  |  |
  Task 6 (Doctor): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 6 (Doctor) | 53.9 (35.86) | 100.0 (75.51) |  |  |
  Task 7 (Word Draw): number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
  Task 7 (Word Draw) | 22.22 (25.06) | 37.55 (25.28) |  |  |
  Task 8 (Typing): number analyzed (Participants) | 10 | 10 | 0 | 0 | 0
  Task 8 (Typing) | 57.7 (61.18) | 73.3 (53.4) |  |  |

19. Secondary Outcome: After-Scenario Questionnaire (ASQ) Score
Description: Aims 1 & 2. The After-Scenario Questionnaire (ASQ) is a 3-item likert-type scale used to assess how difficult a user perceived a task in a usability test. Responses range from 1-strongly disagree to 7- strongly agree. Total score is the sum of the 3 items, possible scores range from 3 to 21. Higher scores indicated better outcomes.
  This was not measured for each task as that was too burdensome for intubated patients. We measured once as an overall rating at the end of the session- 3-item ASQ.
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion
Population: After Scenario Questionnaire is a 3-item patient rating of the usability of the VidaTalk communication application for each communication feature on ease, time, and support information
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 11 | 11 | 0 | 0 | 0
score on a scale
  Task 1 (Tired): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 1 (Tired) | 18.2 (3.92) |  |  |  |
  Task 2 (Pain): number analyzed (Participants) | 11 | 0 | 0 | 0 | 0
  Task 2 (Pain) | 19.5 (2.81) |  |  |  |
  Task 3 (Pain Rating): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 3 (Pain Rating) | 20.3 (1.49) |  |  |  |
  Task 4 (Pain Location): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 4 (Pain Location) | 20.1 (2.02) |  |  |  |
  Task 5 (Pain Quality): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 5 (Pain Quality) | 20.7 (0.949) |  |  |  |
  Task 6 (Doctor): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 6 (Doctor) | 18.1 (4.28) |  |  |  |
  Task 7 (Word Draw): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 7 (Word Draw) | 19.5 (3.81) |  |  |  |
  Task 8 (Typing): number analyzed (Participants) | 10 | 0 | 0 | 0 | 0
  Task 8 (Typing) | 18.1 (5.45) |  |  |  |
  Overall ASQ: number analyzed (Participants) | 0 | 11 | 0 | 0 | 0
  Overall ASQ |  | 17.6 (4.61) |  |  |

20. Secondary Outcome: System Usability Scale (SUS) -Adapted
Description: Aims 1 & 2, System Usability Scale is 13-item likert type scale with item ratings of 1 'strongly agree' to 7 'strongly disagree' to obtain the patient's rating of overall usability of the VidaTalk application, total scores range from 13 to 91
  Note: This is different from the standard 10-item SUS that uses a 5-point scale, with scores ranging 0-100.
Time Frame: Measured during 30-60 minute usability testing visit which occurs at study completion
Population: Note: This is different from the standard 10-item SUS that uses a 5-point scale, with scores ranging 0-100.
  Aim 3 and 5 were not addressed with this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 10 | 11 | 0 | 0 | 0
units on a scale | 82.5 (5.91) | 68.5 (12.37) |  |  |

21. Secondary Outcome: Number of Participants That Responded "Yes" to Having Communication Difficulty at Extubation or ICU Discharge
Description: Measured as a single item : Question asked was - "Presence of communication difficulty in the last few days?" with answers being Yes or No
Time Frame: measured at Extubation /ICU Discharge
Population: Extubated ICU patients
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1- VidaTalk Post-extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention-control | Aim 5-VidaTalk Efficacy in Family Caregivers
Number analyzed (Participants) | 0 | 0 | 22 | 26 | 0
Participants | 0 | 0 | 14 | 23 | 0
Statistical Analysis 1: Comparison: Aim 3 - VidaTalk Tablet App vs Aim 3 - Attention-control; Test type: Superiority; p = 0.05, t-test, 2 sided; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.05 to 1.01]
Statistical Analysis 2: Comparison: Aim 3 - VidaTalk Tablet App; Adjusted for baseline communication difficulty; Test type: Superiority; p = 0.10, Regression, Linear; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.06 to 1.30]

ADVERSE EVENTS:
Time Frame: Aims 1 and 2 - 1 hour observation period Aim 3 - 225 total ICU days for VidaTalk patients. 166 total ICU days for control patients. Average of 8 days for the VidaTalk patients and 6 days for control group. Aim 4 - 10 minute observation period Aim 5 - 6 months post ICU discharge
Description: * All-Cause Mortality: The occurrence of death due to any cause.
  * Serious Adverse Events: Include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions.
  Other (Not Including Serious) Adverse Events: Adverse events that are not Serious Adverse Events.
Groups:
- Aim 1 - VidaTalk Post-Extubation: Specific Aim 1. Develop a commercial prototype of VidaTalk that will include multilingual and customizable messages, compatibility with tablet devices, picture symbols, and integration with mobile communication devices.
- Aim 2 - VidaTalk Intubated: Specific Aim 2. Demonstrate usability with iterative user assessment testing in a clinical setting.
- Aim 3 - VidaTalk Tablet App: Specific Aim 3. Test the clinical efficacy of VidaTalk via android application with MV patients by examining qualitative and quantitative endpoints in a clinical setting. Aim 3 hypothesis: MV patients using VidaTalk will demonstrate significant reductions in patient-reported communication difficulty and frustration, anxiety, sedation exposure, delirium/coma-free days, and improved patient and family satisfaction with ICU care compared to MV patients receiving attention-control (i.e., tablets with health education application).
- Aim 3 - Attention Control: Intubated patients who did not receive the VidaTalk Intervention
- Aim 4: Specific Aim 4. Validation of electronic visual analogue scale, versus current standard paper scale.
- Aim 5 - VidaTalk Efficacy in Family Caregivers - VidaTalk Group: Specific Aim 5 a, b and c. Test the effect of the communication tablet (VidaTalk) on psychological symptoms in family caregivers.
- Aim 5 - Family Caregiver Attention Control: Family members of patients who did not receive the VidaTalk Intervention
- Nurse Focus Group - PreClinical Trial Phase: Focus group of ICU nurses on how to implement the VidaTalk Intervention
- Nurse Focus Group - VidaTalk RCT: Focus group of ICU nurses regarding the utility of the VidaTalk Intervention for communication with patients.
Arm/Group | Aim 1 - VidaTalk Post-Extubation | Aim 2 - VidaTalk Intubated | Aim 3 - VidaTalk Tablet App | Aim 3 - Attention Control | Aim 4 | Aim 5 - VidaTalk Efficacy in Family Caregivers - VidaTalk Group | Aim 5 - Family Caregiver Attention Control | Nurse Focus Group - PreClinical Trial Phase | Nurse Focus Group - VidaTalk RCT
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/23 | 2/31 | 0/32 | 0/0 | 0/18 | 0/16 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/23 | 0/31 | 0/32 | 0/0 | 0/18 | 0/16 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/23 | 0/31 | 0/32 | 0/0 | 0/18 | 0/16 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT02921776/Prot_SAP_002.pdf
  • Informed Consent Form (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02921776/ICF_003.pdf